CLINICAL TRIAL: NCT04164342
Title: Etude de la prévalence de la Douleur Chronique et de Ses Facteurs de Risque après Une Hospitalisation en réanimation Chirurgicale
Brief Title: Prevalence of Chronic Pain and Its Risk Factors After a Surgical Intensive Care Unit Stay. Prospective Observational Cohort
Acronym: DOUCREA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2019-A01865-52
Record Dates: First submitted 2019-11-05; First posted 2019-11-15 (Actual); Last update posted 2022-07-27 (Actual); Status verified 2022-07

CONDITIONS: Pain, Chronic; Critically Ill; Opioid-Related Disorders
Keywords: pain; critically ill
MeSH Terms: conditions — Chronic Pain; Critical Illness; Opioid-Related Disorders; Pain | interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single ARM (Experimental): This is an observational study, all patients will be followed at 3, 6 and 12 months by phone interviews to pass the Brief Pain Inventory (BPI) and the Patient Health Questionnaire-2 (PHQ-2) questionnaires (this is the intervention, since questionnaires at not usually done).
  Interventions: Other: surveys

INTERVENTIONS:
Other: surveys — Phone interviews to pass the Brief Pain Inventory (BPI) and the Patient Health Questionnaire-2 (PHQ-2) questionnaires (this is the intervention, since questionnaires at not usually done) at 3, 6 and 12 months after ICU discharge.

SUMMARY:
The objective of this observational, prospective study is to evaluate the incidence of chronic pain at 3 months after ICU discharge in patients with a prolonged ICU stay (i.e. ≥3 days).

Investigators will assess the proportion of patients with chronic pain (defined according to the Brief Pain Inventory questionnaire), by interview at 3 months after ICU discharge.

All data potentially associated with chronic pain will be collected, including the type of surgery, the acute pain (intensity and duration) during the ICU stay, the type and dose of opioids received, patients comorbidity...

Patients will be follow-up at 6 and 12 months to identify impact on quality of life.

DETAILED DESCRIPTION:
Acute pain is common for ICU patients, with an incidence of 33% at rest and of 56% during nursing care. However, there is few if any data on chronic pain after an ICU stay (ie lasting more than 3 months after ICU discharge), while chronic pain seems to be frequent in patients, in particular following surgeries. Indeed, several studies have shown that in postoperative period, many patients suffer from chronic pains, with incidence from 12 to more than 50 %, depending on surgery.

Known risk factors include:

* Female gender
* young age
* mental disorder antecedent
* pain prior to surgery
* type of anesthesia, including the type and dose of opioids used
* not correctly controlled severe pain
* prolonged pain

Chronic pain is becoming a public health problem, because of its impact on patients quality of life, but also on the over consumption of opioids as a result, and the addiction that arise.

Chronic pain following an ICU stay as been studied so far. Available studies in ICU are mainly interested in the quality of life, which remains altered even many years after ICU discharge. The most popular survey is the SF-36 which includes a section on chronic pain. However no study, to the best of our knowledge, were interested in chronic pain prevalence and in its risk factors after an ICU stay.

In our surgical ICU unit, there is two sedation-analgesia protocols, that use different types of opioids (ie sufentanyl or Remifentanyl), in addition physicians may prescribe morphine for awake patients or other oral opioids. The impact of opioid choice on chronic pain prevalence after ICU discharge is not known today, but could be important, as it is for postoperative chronic pain.

We hypothesis that chronic pain is frequent after a surgical ICU stay and that some factors may be associated with it, including the type of opioids received.

The investigators will conduct a prospective observational study to evaluate this prevalence and the risk factors associated with chronic pain following a prolonged ICU stay.

Patients with an ICU stay ≥3 days, capable to answer to questionnaires will be eligible and will be invited to participate to the study just before their discharge from ICU.

After inclusion, patient's conditions prior to ICU stay, type od admission, all critical care events, pain (duration and intensity), treatments (including opioids)... will be collected.

Investigators will pass the Brief Pain Inventory (BPI) questionnaire A to the patients before discharge from ICU.

Investigators will phone the patient at 3 (primary endpoint), 6 and 12 months after ICU discharge, in order to fill BPI questionnaire for chronic pain diagnosis, to evaluate its impact on quality of life, to fill PHQ 2 survey and record all pain treatment. Beside those 3 phone calls, there is no change in patient care, but patients can be offered to consult their doctor in case of chronic pain screening or presence of depressive symptoms.

This study will allow to characterise chronic pain incidence after an hospitalisation period of at least 3 days in surgical ICU, and to better define possible risk factors. Some risk factors of chronic pain could be modifiable, in particular the type of opioid received. Identification of risk factors for chronic pain could help identifying patients who could benefit from specific care or from post-ICU follow-up consultations.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients
* Hospitalisation in ICU for ≥ 3 days
* Affiliation to French health care coverage
* Oral informed consent of the patient

Exclusion Criteria:

* Patient with chronic pain at inclusion :defined as a prescription of pain killers (level 2 or 3), for more than 3 months
* Cancer with life expectancy < 6 months
* Neurological status not allowing to answer surveys
* Pregnant, nursing or parturient women
* Adult deprived of liberty by court judgment or administrative
* Adult patient protected under the law (guardianship)
* Adult with forced psychiatric care

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2019-11-27 (Actual); Primary Completion 2021-06-25 (Actual); Study Completion 2022-07-26 (Actual)

PRIMARY OUTCOMES:
Proportion of patients suffering from chronic pain 3 months after ICU discharge | 3 months
  Proportion of patients with a Brief Pain Inventory questionnaire positive (answer "YES" at first question) at 3 months after ICU discharge

SECONDARY OUTCOMES:
Proportion of patients suffering from chronic pain at 6 and 12 months after ICU discharge discharge | 12 months
  Proportion of patients with a Brief Pain Inventory questionnaire positive (answer "YES" at first question) 6 and 12 months after ICU discharge
Proportion of patients with possible depressive episode at 3, 6 and 12 months after ICU discharge | 12 months
  Proportion of patients with a score A ≥ 3 ( PHQ-2 score ranges from 0-6). If the score is 3 or greater, major depressive disorder is likely.Patient Health Questionnaire 2 (PHQ 2)

CONTACTS AND LOCATIONS:
Overall Officials: Sigismond SL Lasocki, PU-PH, Study Director — University Hospital, Angers
Locations (1):
- CHU Angers, Angers, France